CLINICAL TRIAL: NCT04748055
Title: A Pilot Study Examining Changes in Nasal IL-1 During Acute Asthma Exacerbation in Adolescents
Brief Title: Examining Changes in Nasal IL-1 During Acute Asthma Exacerbation in Adolescents
Acronym: Attack Asthma
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 20-2452; R01HL135235 (NIH)
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2023-10

CONDITIONS: Asthma
Keywords: Asthma in children; Asthma attack
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — NELF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To study the change from baseline in IL-1β (interleukin 1 beta) concentrations in the nasal airway during acute asthma exacerbation, specifically to measure the degree of change and identify the timing of peak IL-1β concentration. This information will allow the investigators to estimate effect size and guide decisions about the optimal timing of anakinra administration for the future study.

DETAILED DESCRIPTION:
The study team will recruit 60 teens and young adults with persistent asthma who are at high risk for future exacerbation from the University of North Carolina at Chapel Hill (UNC) Children's Allergy and Asthma Center in Raleigh, NC. Participants will complete 13 study visits: an initial in-person visit (the study team will make every attempt to coordinate this visit with a scheduled clinic visit) and 12 monthly virtual follow up visits. Participants will be asked to use an at home spirometer once daily in the evening and will also complete an electronic asthma survey each night. Participants will also be provided with a sensor that tracks their rescue medication use throughout the study. Participants will undergo collection of nasal epithelial lining fluid (NELF) at the baseline visit. During the 12 months of study, participants will self-collect NELF samples if certain prespecified criteria for asthma exacerbation are met. Samples will be analyzed for IL-1β, interleukin receptor antagonist (IL-1RA) and other mediators associated with acute asthma exacerbation. Virtual follow up visits using a video platform will occur monthly for 12 months. Participants will self-report healthcare utilization and prescription for systemic corticosteroids. Spirometry and symptom survey data will be matched to subject-reported asthma exacerbations. The study design is adapted to minimize in-person visits, using web-based platforms for virtual visits and self-collection of samples to prioritize safety during the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Ages 12 to 21 years, inclusive, of both genders
* Physician diagnosis of persistent asthma or symptoms consistent with persistent asthma based on expert guidelines for diagnosis and management of asthma (1).
* Current use of a controller therapy such as an inhaled corticosteroid (ICS), ICS in combination with long-acting beta agonist (LABA), or leukotriene receptor antagonist (LTRA).
* Asthma is "not well controlled" (participant must have ≥1 of the following):

  * Asthma Control Test (ACT) score <20,
  * FEV1 <80% of predicted,
  * Meets Global Initiative on Asthma (GINA) criteria for partly controlled or uncontrolled asthma (2):

In the past 4 weeks, has the patient had:

* Daytime symptoms >2x/week?
* Any night waking due to asthma?
* SABA reliever needed >2x/week?
* Any activity limitation due to asthma?

  * [0 = Well controlled; 1-2 = Partly controlled; 3-4 = Uncontrolled]
  * A history of at least one exacerbation requiring systemic corticosteroids (oral, IM or IV) in the past 24 months

    * Access to a smartphone
    * Wireless internet access in the participant's home
    * Access to a standard freezer in the home

Exclusion Criteria:

* Systemic corticosteroid-dependent asthma (i.e. people who take oral steroids such as prednisone daily for asthma control). Use of other immunomodulator medications (such as biologics for asthma like omalizumab, etc) is allowable so long as the participant has been on a stable dose of the medication for at least 3 months.
* Participants whose asthma is sufficiently severe that the participants routinely require rescue albuterol multiple times a day for symptom relief (not including pre-exercise albuterol use).
* Pulmonary disease other than asthma that in the opinion of investigators may affect the interpretation of spirometry data, including but not limited to vocal cord dysfunction, restrictive lung disease, or cystic fibrosis.
* Inability to perform spirometry.
* History of spirometry-induced bronchoconstriction.
* Pregnancy or nursing a baby. Due to the effect of hormonal changes of pregnancy/lactation on airway inflammation, participants who are pregnant or nursing will be excluded from study.

Ages: 12 Years to 21 Years | Sex: All
Age Groups: Child, Adult
Study Population: The study team will recruit 60 teens and young adults with persistent asthma who are at high risk for future exacerbation from the UNC Children's Allergy and Asthma Center in Raleigh, NC.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Nasal IL-1β (pg/mL) Concentrations over time during Asthma Exacerbation | Baseline and up to 5 days from the time asthma exacerbation is diagnosed
  Nasal epithelial lining fluid (NELF) is collected during a period of wellness (baseline) and daily during acute asthma exacerbation (defined by pre-specified criteria) for 5 days. The change from baseline in nasal IL-1β concentrations during acute asthma exacerbation will be measured for each of the 5 days of the exacerbation to measure the degree of change over time and to identify the timing of peak IL-1β concentration.

SECONDARY OUTCOMES:
Change from Baseline in Forced Expiratory Volume in the First Second (FEV1) Percent (%) Predicted over time during Asthma Exacerbation | Baseline and up to 5 days from the time asthma exacerbation is diagnosed
  FEV1 will be measured during a period of wellness (baseline) and daily during acute asthma exacerbation defined by pre-specified criteria for 5 days. The change from baseline in FEV1 % predicted during asthma exacerbation will be measured for each of the 5 days of the exacerbation to determine the degree of change over time.
Change from Baseline in Nasal Concentrations of Other Relevant Inflammatory Cytokines/Chemokines over time during Asthma Exacerbation | Baseline and up to 5 days from the time asthma exacerbation is diagnosed
  Nasal epithelial lining fluid (NELF) is collected during a period of wellness (baseline) and daily during acute asthma exacerbation defined by pre-specified criteria for 5 days. The change from baseline in nasal cytokine and chemokine concentrations during acute asthma exacerbation will be measured for each of the 5 days of the exacerbation to determine the degree of change over time.
Correlation over time Between Changes in Nasal IL-1β Concentration from Baseline and Changes in FEV1 % Predicted from Baseline during Asthma Exacerbation | Baseline and up to 5 days from the time asthma exacerbation is diagnosed
  Assess the relationship over time between the asthma exacerbation-induced change in NELF IL-1β concentrations and the asthma exacerbation-induced change in FEV1% predicted. The correlation will be calculated for each of the 5 days of the exacerbation to determine the degree of change over time.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Burbank, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: 9 to 36 months following publication
Access Criteria: Approved IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] National Asthma Education and Prevention Program. Expert Panel Report 3 (EPR-3): Guidelines for the Diagnosis and Management of Asthma-Summary Report 2007. J Allergy Clin Immunol. 2007 Nov;120(5 Suppl):S94-138. doi: 10.1016/j.jaci.2007.09.043. PMID 17983880